CLINICAL TRIAL: NCT07087171
Title: Assessing the Impact of an Artificial Intelligence-Machine Learning Model on Patient Engagement in Medically Assisted Reproduction
Brief Title: AI-Driven Model Impact on Patient Engagement in Medically Assisted Reproduction
Status: Recruiting | Type: Observational
Sponsor: Instituto Valenciano de Infertilidade de Lisboa (Network)
Collaborators: Univfy Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2412-LIS-233-AN
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Infertility (IVF Patients); Artificial Intelligence (AI)
Keywords: IVF; Artificial intelligence; counselling; Conversion rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional counselling group: A retrospective cohort of patients who underwent their new patient visit with one of the doctors participating in the study between December 2024 and June 2025 will be analyzed.
- AI-based counselling group: A prospective cohort of patients undergoing their NPV with one of the doctors participating in the study will receive an artificial intelligence-machine learning report with their accurate personalized probabilities of having a live birth rate together with a medical explanation by their physician
  Interventions: Other: Artificial intelligence-Machine learning report with accurate personalized probabilities of having a live birth rate

INTERVENTIONS:
Other: Artificial intelligence-Machine learning report with accurate personalized probabilities of having a live birth rate — Patients included in the prospective arm will receive the Univfy® PreIVF Report with their accurate personalized probabilities of having a live birth rate (Univfy®) together with a medical explanation by their physician
  Groups: AI-based counselling group

SUMMARY:
Infertility is a globally significant medical condition, profoundly impacting individuals and couples both emotionally and physically. The multifaceted nature of in vitro fertilization (IVF) treatment demands active patient participation, with engagement playing a pivotal role in treatment success and satisfaction. However, suboptimal engagement can lead to challenges such as not initiating treatment, missed appointments, medication errors, dropping out and heightened stress levels, all of which may adversely affect clinical outcomes.

Recent advancements in Artificial Intelligence (AI) and Machine Learning (ML) have revolutionized healthcare, offering innovative solutions for personalized patient care. In IVF, AI-ML models hold the potential to enhance patient engagement by delivering tailored communication, reminders, and educational support, but also improved prognostication by providing personalized and accurate predictions of treatment outcomes. These capabilities enable patients to make more informed decisions and enhance their adherence to treatment protocols.This protocol outlines a prospective evaluation of an AI-ML model, specifically the Univfy PreIVF report, developed to improve patient engagement in IVF care. Recently, a retrospective, multicenter study reported improved IVF utilization rates among patients counselled using the Univfy PreIVF Report. The current study will prospectively assess the model's effectiveness in addressing individual patient needs and creating a supportive treatment environment. Specifically, this study will measure adherence to providers' recommendation of treatment protocols. By analyzing the impact of these interventions, this research aims to provide robust evidence for the integration of AI-ML technologies in reproductive medicine, paving the way for broader implementation and improved patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Infertile patients aged 18-45 years
* Patients willing to undergo Medically Assisted Reproduction (heterosexual couples, same-sex female couples and single females undergoing artificial insemination, IVF/ICSI or oocyte donation treatments)

Exclusion Criteria:

* Age >45 years
* Patients who are not candidates for IVF/ICSI
* Patients who are menopausal or peri-menopausal
* Patients undergoing Fertility Preservation
* Same-sex couples who will undergo reception of oocytes from partner.
* Patients who decline to be counselled about their probability of having a live birth from IVF/ICSI treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study period will run from December 1, 2024, to December 31, 2025. During the first phase, from December 1, 2024, to May 31, 2025, a retrospective cohort of patients attending their first appointment at IVI Lisboa with a research team member will have received conventional counseling regarding IVF treatment prognosis. In the second phase, from June 1, 2025, to November 30, 2025, a prospective cohort of patients attending their first appointment with the same team will receive AI-based counseling using the Univfy® PreIVF Report.®.
Sampling Method: Non-Probability Sample
Enrollment: 774 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
9-month conversion rate | From enrollment until 9 months after
  9-month conversion, with conversion being defined as the first usage of Medically Assisted Reproduction (MAR) following a new patient visit

SECONDARY OUTCOMES:
3-month MAR conversion | From enrollment until 3 months after
  3-month conversion rate
6-month MAR conversion | From enrollment until 6 month after
  6-month conversion

CONTACTS AND LOCATIONS:
Locations (1):
- IVI-RMA Lisboa, Lisbon, Portugal